CLINICAL TRIAL: NCT06410118
Title: Efficacy of the DreamChanger Intervention in Combination With Imagery Rehearsal Therapy to Reduce Nightmares in Children
Brief Title: The DreamChanger Intervention in Combination With Imagery Rehearsal Therapy for Children's Nightmares
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Michal Kahn, Senior lecturer, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0008185-1
Record Dates: First submitted 2024-05-05; First posted 2024-05-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Nightmare

STUDY DESIGN:
Intervention Model Description: The intervention group will be compared to a waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DreamChanger combined with Imagery Rehearsal Therapy (Experimental): Families will receive the DreamChanger remote along with 3 instructional videos for parents, explaining how to present the remote to children, and how to rehearse alternative dream imagery using the DreamChanger remote.
  Interventions: Behavioral: DreamChanger+IRT
- Waitlist control (No Intervention): Families will be placed on a waitlist, and receive the intervention 6 weeks after baseline

INTERVENTIONS:
Behavioral: DreamChanger+IRT — Families will receive the DreamChanger remote along with 3 instructional videos for parents, explaining how to present the remote to children, and how to rehearse alternative dream imagery using the DreamChanger remote.
  Arms: DreamChanger combined with Imagery Rehearsal Therapy

SUMMARY:
This clinical trial will test the efficacy of parent-delivered DreamChanger Intervention in combination with Imagery Rehearsal Therapy (IRT) for reducing the frequency and severity of nightmares in children aged 3-10. Children will be randoimized to either the combined intervention or to a waitlist control group.The intervention will include providing children with the DreamChanger remote, and providing parents with instructional videos, explaining how to use the device along with the IRT strategy to address nightmares.

At baseline, mid-treatment, and post-treatment, parents in both groups will complete questionnaires asking about the child's nightmares, sleep, externalizing and internalizing symptoms, PTSD symptoms, demographic characteristics, and parent sleep and distress. Parents in the intervention group will also be asked to complete questionnaires regarding their compliance and satisfaction with the intervention, as well as a 3-month follow-up assessment.

DETAILED DESCRIPTION:
Nightmares, characterized as distressing dreams often leading to awakening, are relatively common in young children. However, approximately 3-6% of children endure recurrent nightmares, occurring at least once per week, causing significant distress and impairment. These persistent nightmares can be idiopathic or post-traumatic, and may be linked to conditions such as nightmare disorder or post-traumatic stress disorder (PTSD). Children experiencing recurrent nightmares face an elevated risk for various maladaptive consequences, including reduced sleep quality and quantity, heightened nocturnal anxiety, and challenges in emotional, social, and academic functioning. Moreover, parents often experience disruptions in their own sleep, which may lead to adverse health outcomes. Hence, the demand for effective interventions to mitigate the multifaceted burdens associated with recurrent nightmares is pronounced.

The most established intervention for children struggling with recurrent nightmares is Imagery Rehearsal Therapy (IRT). This approach aims to diminish the frequency and intensity of nightmares by encouraging children to engage with and modify the content of their nightmares through visualization and rehearsal techniques. Studies assessing the efficacy of IRT in children have demonstrated significant reductions in nightmare frequency and associated distress following treatment. However, the evidence base for this intervention remains limited, with only one small-scale (N=20) randomized controlled trial (RCT) conducted in children to date. Correspondingly, there is a critical need for further research to evaluate treatment effectiveness in children.

Furthermore, despite the promise of IRT in reducing nightmare frequency and intensity, approximately 30% of children do not sufficiently benefit from treatment. This underscores the necessity to refine and tailor this intervention to better address the characteristics of children. To date, research has yet to explore the potential advantages of augmenting IRT with additional components. The DreamChanger intervention offers a novel approach specifically designed for young children experiencing recurrent nightmares. Utilizing a remote-control-like device emitting a soft light, this cognitive intervention empowers children to "change the channel of their dreams", fostering a sense of mastery and control. A recent RCT demonstrated the efficacy of the DreamChanger in reducing nightmares and anxiety in young children. Building upon these findings, we posit that combining IRT with the DreamChanger may enhance treatment outcomes. Encouraging children to utilize the DreamChanger remote during the rehearsal of alternative dream scenarios may establish associations between the remote and alternative dream imagery, potentially improving the mental accessibility of imagery when using the remote at night. Thus, the DreamChanger has the potential to augment IRT by further stimulating the child's imagination and sense of mastery, while also facilitating the rehearsal and accessibility of alternative dream imagery.

This study seeks to advance scientific knowledge regarding interventions for pediatric nightmares by examining the efficacy of a novel treatment approach - a combination of IRT with the DreamChanger intervention - to alleviate recurrent nightmares and improve sleep quality in young children. This augmented intervention will be compared to a waitlist control group in an RCT. The research plan is based on an RCT design, with 2 arms (intervention vs waitlist control) and assessment points at baseline, mid-treatment, post-treatment, and for the intervention group - an additional 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* child aged 3-10 years
* parents aged over 18 years
* child experiencing distressing nightmares at least once per week on average, for at least 1 month.

Exclusion Criteria:

* Child receiving concurrent treatment for nightmares, sleep, or anxiety
* Child diagnosed with a medical sleep problem (e.g., OSA, RLS)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Nightmare frequency and severity | Baseline, mid-treatment (2 weeks following baseline), post-treatment (4 weeks following baseline), and at a 3-month follow up
  Nightmare severity, frequency and related distress, as assessed using a modified version of the Nightmare Disorder Index

SECONDARY OUTCOMES:
Child sleep problems | Baseline, mid-treatment (2 weeks following baseline), post-treatment (4 weeks following baseline), and at a 3-month follow up
  Sleep difficulties such as frequent awakenings, prolonged nighttime wakefulness, and short sleep duration, as assessed uding the Child Sleep Habits Questionnaire.
Child externalizing and internalizing problems | Baseline, post-treatment (4 weeks following baseline), and at a 3-month follow up
  Child behavioral problems, as assessed using the Strengths and Difficulties Questionnaire
Parent distress | Baseline, post-treatment (4 weeks following baseline), and at a 3-month follow up
  Parent depression, anxiety, and stress symptoms, as assessed using the DASS-21.

OTHER OUTCOMES:
Parent compliance and satisfaction with the intervention | Mid-treatment and post-treatment (4 weeks following baseline)
  Parent adherence to the intervention (e.g., watching the instructional videos, rehearsing the alternative dream scenarios, etc.) will be assessed, along with items regarding parents' satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kahn, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No